CLINICAL TRIAL: NCT00787384
Title: Therapeutic and Biological Effects of Imatinib Mesylate in Primary Hypereosinophilic Syndromes
Brief Title: Efficacy of Imatinib Mesylate in Hypereosinophilic Syndromes
Acronym: NILG-HES1-03
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Responsible Party: Dr Renato Bassan, NILG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NILG-HES1-03; EUDRACT 2004-002280-24
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-12

CONDITIONS: Hypereosinophilic Syndrome; Chronic Eosinophilic Leukemia; Chronic Idiopathic Hypereosinophilia
Keywords: Hypereosinophilic syndrome (HES); chronic eosinophilic leukaemia (CEL); chronic idiopathic hypereosinophilia (CIH); Imatinib; Response; Timing to response
MeSH Terms: conditions — Hypereosinophilic Syndrome; Pdgfra-Associated Chronic Eosinophilic Leukemia | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib (Experimental): Patients received oral imatinib 100 mg/d; in case of unsatisfactory response (less than complete) Imatinib could be increased by 100 mg/die on a weekly basis and up to a maximum of 400 mg/die. Imatinib was discontinued after 12 total weeks of therapy.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Patients received oral imatinib 100 mg/d; in case of unsatisfactory response (less than complete) Imatinib could be increased by 100 mg/die on a weekly basis and up to a maximum of 400 mg/die. Imatinib wsa discontinued after 12 total weeks of therapy.
  Other Names: Gleevec

SUMMARY:
The study was performed to assess: 1) clinical activity of Imatinib in patients with HES, CEL and CIH; 2) correlation between Imatinib activity and specific disease subtype; 3) long-term outcome of HES, CEL and CIH patients treated with Imatinib; 4) safety and tolerability of Imatinib administration.

DETAILED DESCRIPTION:
Hypereosinophilic syndrome (HES), chronic eosinophilic leukaemia (CEL) and chronic idiopathic hypereosinophilia (CIH) are rare disorders characterized by chronic hypereosinophilia with possible damage to various organs due to eosinophilic infiltration and release of cytokines. The therapies of these diseases are largely unsatisfactory and based on the use of a variety of antiproliferative drugs such as corticosteroids, interferon-alfa, cyclosporine, vincristine or hydroxyurea. More often the responses are transient and patients need numerous treatment lines.

In 2001 Schaller et al reported the first case of a patient with HES resistant to conventional treatment that responded to imatinib mesylate. (Schaller, MGM 2001). After that, many authors described cases with hypereosinophilia that achieve a rapid response to Imatinib and in 2003 Cools et al identified a novel tyrosine kinase generated from the fusion of the Fip1-like 1 (FIP1L1) gene to the PDGFRalfa gene associated to hypereosinophilia.

The optimal dose of Imatinib in this setting of patients is still unknown; however, the demonstration of effective and safe clinical doses in a variety of currently studied malignant diseases, suggests that a dose of 100 mg/day increasing weekly of 100 mg/day (maximum dose 400 mg/day), may be employed.

We designed a phase II trial to investigate the clinical anti-proliferative activity, safety and tolerability of escalating doses of Imatinib (entry dose 100 mg/d)administered for 12 total weeks in HES, CEL and CIH patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of HES, CEL and CIH, who are either previously untreated or have been treated with corticosteroids, cytotoxic drugs, and IFN.
* age > 15 years.
* signature of a written informed consent(by parents/tutors for patients aged < 18 years).

Exclusion Criteria:

* patients with a diagnosis of secondary hypereosinophilia
* age < 15 years

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Safety: Adverse events and serious adverse events
Time to response
Diagnostic profile of Imatinib-responsive cases
Duration of responses following drug withdrawal after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, MD, Principal Investigator — USC Ematologia Ospedali Riuniti di Bergamo
Locations (4):
- Italy (4):
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo, Bergamo
  - Divisione di Ematologia Spedali Civili di Brescia, Brescia, Brescia
  - USC Ematologia Azienda Ospedaliera Università Careggi, Florence, Firenze
  - UO Ematologia, Azienda Ospedaliera ULSS6, Vicenza, Vicenza

REFERENCES:
- [Result] Intermesoli T, Delaini F, Acerboni S, Salmoiraghi S, Spinelli O, Guerini V, Vannucchi AM, Mappa S, Rossi G, Rossi V, Di Bona E, Paratore S, Carobbio A, Rambaldi A, Barbui T, Bassan R. A short low-dose imatinib trial allows rapid identification of responsive patients in hypereosinophilic syndromes. Br J Haematol. 2009 Dec;147(5):681-5. doi: 10.1111/j.1365-2141.2009.07893.x. Epub 2009 Sep 4. PMID 19735261